CLINICAL TRIAL: NCT00127478
Title: A Phase II/III Extension Study to Evaluate the Safety and Tolerability of Atrasentan
Brief Title: A Long Term Safety Study With Atrasentan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M01-304
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Prostate Cancer; Adenocarcinoma
Keywords: Hormone Refractory Prostate Cancer; Adenocarcinoma of the Prostate
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Atrasentan

INTERVENTIONS:
Drug: Atrasentan

SUMMARY:
The primary purpose of the study is to evaluate long-term safety and tolerability of atrasentan 10 mg in men with hormone refractory prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years, inclusive;
* Subject is currently active in an atrasentan clinical study OR has histologically or cytologically documented diagnosis of prostate adenocarcinoma and is considered hormone refractory;
* Karnofsky Performance Score greater than or equal to 60;
* Adequate hematologic function and liver function tests;
* No New York Heart Association (NYHA) class greater than or equal to 2.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2001-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Adverse events | Every 12 weeks
Serious adverse events
Oncology-related events (OREs)
Deaths
Study drug exposure
Change from baseline in Karnofsky performance status
Vital signs
Stratification by treatment group from prior study

SECONDARY OUTCOMES:
Safety and laboratory parameters | Every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary Gordon, MD, Study Director — Abbott
Locations (15):
- United States (7):
  - Prostate Oncology Specialists, Marina del Rey, California
  - Western Clinical Research, Inc., Torrance, California
  - South Florida Medical Research, Aventura, Florida
  - Beth Isreal Medical Center, Phillips Ambulatory Care Ceneter, New York, New York
  - ViaHealth Rochester General Hospital Center for Urology, Rochester, New York
  - Oregon Urology Specialist, Division of Clinical Research, Springfield, Oregon
  - University of Pittsburgh Department of Urology, Pittsburgh, Pennsylvania
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - CroMedia Prime/Prime Trials Vancouver Hospital, Vancouver, British Columbia
  - Ken Janz MD, Burlington, Ontario
  - McMaster Institute of Urology, Hamilton, Ontario
  - McGill University Health Center Royal VIctoria Hosptial, Montreal, Quebec
- Hoptial de Ranguell Service d'Urologie, Toulouse, Cedex, France
- University Hospital Rotterdam, Department of Urology, Rotterdam, Netherlands
- Leighton Hospital Urology Research Dept., Michael Heal Outpatients Dept., Crewe, United Kingdom